CLINICAL TRIAL: NCT03160820
Title: Comparison of Immunization Schedules of Beijing Tiantan Biological's MMR Vaccine in 18-72 Month-Old Children
Brief Title: Study on Immunization Schedule of Beijing Tiantan Biological's Measles-mumps-rubella(MMR) Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Beijing Tiantan Biological Products Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wu Jiang, Director of Department of Immunization and Prevention,Beijing Center for Disease Control and Prevention. Principal Investigator, Public Health Chief Physician, Centers for Disease Control and Prevention, China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BJCDCWJ201601
Record Dates: First submitted 2017-05-10; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Measles; Mumps; Rubella; Adverse Event Following Immunisation
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- one dose of MMR (Other): Subjects are vaccinated with MMR(Measles, mumps and rubella Combined Vaccine, Live) on 18 months old.
  Interventions: Biological: Measles, mumps and rubella Combined Vaccine, Live
- 30 months after two doses of MMR (Other): Subjects are vaccinated two doses of MMR(Measles, mumps and rubella Combined Vaccine, Live) on 18 month and 4 years old, sequentially.
  Interventions: Biological: Measles, mumps and rubella Combined Vaccine, Live
- 42 months after two doses of MMR (Other): Subjects are vaccinated two doses of MMR(Measles, mumps and rubella Combined Vaccine, Live) on 18 month and 5 years old, sequentially.
  Interventions: Biological: Measles, mumps and rubella Combined Vaccine, Live
- 54 months after two doses of MMR (Other): Subjects are vaccinated two doses of MMR(Measles, mumps and rubella Combined Vaccine, Live) on 18 month and 6 years old, sequentially.
  Interventions: Biological: Measles, mumps and rubella Combined Vaccine, Live

INTERVENTIONS:
Biological: Measles, mumps and rubella Combined Vaccine, Live — Subjects will be inoculated one dose of MMR vaccine and collected blood samples before and after vaccination.
  Other Names: Beijing Tiantan Biological Products Co., Ltd

SUMMARY:
This study will evaluate the immunogenicity and safety of Beijing Tiantan's MMR vaccine in subjects 18 months of age and older. The MMR vaccine may be administered as a second dose to 4-6 year-old persons with one dose immunization with MMR vaccine or as a first dose to 18 month-old subjects with one dose immunization with measles-rubella(MR).

DETAILED DESCRIPTION:
This study will evaluate the immunogenicity and safety of Beijing Tiantan's MMR vaccine in subjects 18 months of age and older.

The MMR vaccine may be administered as a second dose to 4-6 year-old persons with one dose immunization with MMR vaccine or as a first dose to 18 month-old subjects with one dose immunization with MR.

Immune efficacy and safety will be compared among different immunization schedules,including inoculation doses,enhanced immunity age,vaccination interval time.

Antibody persistence of 1 dose of MMR vaccine will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy children; 150 subjects 18 months old; 150 subjects 4 years old;300 subjects 5 years old; 150 subjects 6 years old; their guardians signed informed consent;
* undiagnosed as measles, mumps and rubella;
* in good health as determined by the outcome of medical history, physical examination and clinical judgment; suitable to MMR immunization;
* guardians would comply with the requirements of the protocol;
* immunized with MR or measles vaccine(MV) at 8 months old;immunized with MMR at 18 months old(not applicable to subjects 18 months old); unvaccinated by biological products within one month;
* Axillary temperature ≤37℃;
* the local household population or permanent population;

Exclusion Criteria:

* history of allergic disease or reactions likely to be exacerbated by any component of the vaccine(any previous vaccination history of allergies and egg allergy history);
* Current confirmed as acute disease, severe chronic diseases or acute development of chronic diseases;
* Participating in another clinical trial at the same time;

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 873 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the MMR vaccines in terms of antibody concentration | through study completion, an average of 1 year
  For measles virus, seroresponse is defined as post-vaccination anti-measles virus antibody concentration (Ab conc) >200 mIU/mL.
  For mumps virus, seroresponse is defined as post-vaccination anti-mumps virus Ab conc >100 IU/mL.
  For rubella virus, seroresponse is defined as post-vaccination anti-rubella virus Ab conc >20 IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Principal Investigator — Beijing Center for Diseases Control and Prevention
Locations (4):
- China (4):
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Inner Mongolia Center for Disease Control and Prevention, Hohhot, Inner Mongolia
  - Shanxi Provincial Center for Disease Control and Prevention, Taiyuan, Shanxi
  - Tianjin Center for Disease Control and Prevention, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No